CLINICAL TRIAL: NCT01574768
Title: LATERAL PHARYNGOPLASTY OUTCOMES IN THE TREATMENT OF SNORE AND OBSTRUCTIVE SLEEP APNEA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital do Servidor Publico Estadual (Other)
Collaborators: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, CAROLINA DE ANDRADE FERREIRA VIEIRA, otolaryngologist, Hospital do Servidor Publico Estadual
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 135/11
Record Dates: First submitted 2012-04-07; First posted 2012-04-10 (Estimated); Last update posted 2012-04-10 (Estimated); Status verified 2012-04

CONDITIONS: Snore; Obstructive Sleep Apnea
MeSH Terms: conditions — Snoring; Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Lateral Pharyngoplasty — Tonsilectomy, microdissection of the superior pharyngeal constrictor muscle within the tonsillar fossa and sectioning of this muscle

SUMMARY:
The aim of this study is to describe the results of Lateral Pharyngoplasty in the treatment of snore and OSAS.

ELIGIBILITY:
Inclusion Criteria:

* snore
* osas

Exclusion Criteria:

* previous pharynx surgery
* use of medication that modifies the muscular tonus or the perception of sleepiness before or after the surgery
* body mass index (BMI) bigger than 35 kg/m2
* neurological or psychiatric disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2011-11; Primary Completion 2012-08 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
AHI | 6 months
  Change in AHI

CONTACTS AND LOCATIONS:
Overall Officials: Michel B Cahali, MD, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- Hospital do Servidor Público Estadual, São Paulo, São Paulo, Brazil